CLINICAL TRIAL: NCT03988465
Title: HemoSonics - UTMB Cardiac Surgery Study
Status: Completed | Type: Observational
Sponsor: HemoSonics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HEMCS-024
Record Dates: First submitted 2019-06-10; First posted 2019-06-17 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Blood Loss, Surgical
Keywords: Viscoelastic testing; Coagulation; Quantra; Hemostasis
MeSH Terms: conditions — Blood Loss, Surgical; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Cardiac Surgery Patients: Patients undergoing cardiopulmonary bypass surgery, including placement of a ventricular access device.
  Interventions: Diagnostic Test: Quantra System

INTERVENTIONS:
Diagnostic Test: Quantra System — Diagnostic device to monitor coagulation properties of a whole blood sample at the point-of-care.
  Other Names: Quantra QPlus Cartridge

SUMMARY:
This study will evaluate the performance of the Quantra System comprised of the Quantra Hemostasis Analyzer with the Quantra QPlus Cartridge in patients undergoing cardiac surgery utilizing cardiopulmonary bypass, including the placement of a ventricular access device.

DETAILED DESCRIPTION:
The Quantra System is a fully integrated and automated in vitro diagnostic device which uses SEER Sonorheometry, and ultrasound-based technology, to characterize the viscoelastic properties of a whole blood sample during coagulation. The Quantra QPlus Cartridge was developed to monitor hemostasis during major surgical procedures in adult patients. The cartridge consists of four independent channels each containing different sets of reagents, which provide four measurements performed in parallel yielding six parameters that depict the functional status of a patient's coagulation system.

This single-center, prospective, observational study will evaluate the performance of the Quantra System as compared to and comparable measures determined using the TEG 5000.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years
* Subject is scheduled for cardiac surgery utilizing cardiopulmonary bypass, including the placement of a ventricular access device.
* Subject is willing to participate, and he/she has signed a consent form.

Exclusion Criteria:

* Subject is younger than 18 years
* Subject is unable to provide written informed consent
* Subject is incarcerated at the time of the study
* Subject is pregnant
* Subject is currently enrolled in a distinct study that might confound the results of the proposed study
* Subject is affected by a condition that, in the opinion of the clinical team, may pose additional risks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes subjects 18 years or older undergoing cardiac surgery utilizing cardiopulmonary bypass, including placement of a ventricular access device.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Comparison of Quantra Clot Time results to TEG R results | Baseline, defined as after induction of anesthesia but before surgical incision
  Coagulation function assessed by Quantra and TEG 5000
Comparison of Quantra Clot Stiffness results to TEG MA results | Baseline, defined as after induction of anesthesia but before surgical incision
  Coagulation function assessed by Quantra and TEG 5000
Comparison of Quantra Clot Time results to TEG R results | During bypass
  Coagulation function assessed by Quantra and TEG 5000
Comparison of Quantra Clot Stiffness results to TEG MA results | During bypass
  Coagulation function assessed by Quantra and TEG 5000
Comparison of Quantra Clot Time results to TEG R results | Post-bypass, defined as 10 to 20 minutes after protamine administration
  Coagulation function assessed by Quantra and TEG 5000
Comparison of Quantra Clot Stiffness results to TEG MA results | Post-bypass, defined as 10 to 20 minutes after protamine administration
  Coagulation function assessed by Quantra and TEG 5000
Comparison of Quantra Clot Time results to standard coagulation test results (aPTT) | Baseline, defined as after induction of anesthesia but before surgical incision
  Coagulation function assessed by Quantra and standard coagulation tests
Comparison of Quantra Clot Stiffness results to laboratory fibrinogen results | Baseline, defined as after induction of anesthesia but before surgical incision
  Coagulation function assessed by Quantra and standard coagulation tests
Comparison of Quantra Clot Stiffness results to laboratory-determined platelet count | Baseline, defined as after induction of anesthesia but before surgical incision
  Coagulation function assessed by Quantra and standard coagulation tests
Comparison of Quantra Clot Time results to standard coagulation test results (aPTT) | During bypass
  Coagulation function assessed by Quantra and standard coagulation tests
Comparison of Quantra Clot Stiffness results to laboratory fibrinogen results | During bypass
  Coagulation function assessed by Quantra and standard coagulation tests
Comparison of Quantra Clot Stiffness results to laboratory-determined platelet count | During bypass
  Coagulation function assessed by Quantra and standard coagulation tests
Comparison of Quantra Clot Time results to standard coagulation test results (aPTT) | Post-bypass, defined as 10 to 20 minutes after protamine administration
  Coagulation function assessed by Quantra and standard coagulation tests
Comparison of Quantra Clot Stiffness results to laboratory fibrinogen results | Post-bypass, 10 to 20 minutes after protamine
  Coagulation function assessed by Quantra and standard coagulation tests
Comparison of Quantra Clot Stiffness results to laboratory-determined platelet count | Post-bypass, defined as 10 to 20 minutes after protamine administration
  Coagulation function assessed by Quantra and standard coagulation tests

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No